CLINICAL TRIAL: NCT06111326
Title: A Phase Ib/II Clinical Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of BC3402 in Combination With Durvalumab in Patients With Advanced Hepatocellular Carcinoma
Brief Title: BC3402 in Combination With Durvalumab in Patients With Advanced Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biocity Biopharmaceutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC3402-105
Record Dates: First submitted 2023-10-17; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BC3402+Durvalumab (Experimental): Subjects will receive BC3402 and Durvalumab in a treatment cycle.
  Interventions: Drug: BC3402 injection; Drug: Durvalumab injection

INTERVENTIONS:
Drug: BC3402 injection — Intravenous infusion, once every 2 weeks, 4 weeks/cycle.
Drug: Durvalumab injection — Intravenous infusion, once every 4 weeks, 4 weeks/cycle.

SUMMARY:
Phase Ib: Dose exploration: To assess the safety, tolerability, and determine the recommended Phase 2 dose (RP2D) of BC3402 in combination with durvalumab in subjects with advanced hepatocellular carcinoma (HCC) Phase II: Dose Expansion: To assess the antitumor activity of BC3402 in combination with durvalumab in subjects with advanced HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to participate in the study and sign an informed consent form;
2. Male or female aged ≥ 18 years and ≤ 75 years;
3. Patients with advanced hepatocellular carcinoma confirmed by histology or cytology, or cirrhosis which meets the clinical diagnostic criteria of hepatocellular carcinoma by the by American Association for the Study of Liver Disease (AASLD) (2018 edition);
4. ECOG performance status of 0 or 1;
5. HBV Patients with HBV infection must be treated with antiviral therapy to ensure adequate viral suppression prior to enrollment;
6. Adequate organ and marrow function;
7. Male or female subjects with childbearing potential must agree to use reliable contraceptive methods.

Exclusion Criteria:

1. Received local hepatic therapy within 4 weeks prior to initiation of the study drug;
2. History of hepatic encephalopathy within the past 12 months or a requirement for medications to prevent or control encephalopathy;
3. The subject has clinically significant ascites requiring therapeuticc peritonrocentesis or peritoneal drainage.
4. The subject has main portal vein thrombosis on baseline imaging;
5. Documented history of GI bleeding within the past 6 months or at a high risk of GI bleeding per the investigator's clinical judgement;
6. Current or prior use of systemic corticosteroids or other immunosuppressive agents within 2 weeks before initiation of study drug;
7. Prior treatment with any anti-TIM3 antibody;
8. Prior treatment with an anti-PD-1 or anti PD-L1 immune checkpoint inhibitor antibody (only applicable for dose expansion part).

Other protocol-defined Inclusion/Exclusion may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Phase Ib: Dose Exploration Part-The incidence of dose limiting toxicity (DLT) events | 28 Days
  To assess the incidence of dose limiting toxicity (DLT) events at different doses of BC3402 in combination with durvalumab in the treatment of advanced HCC
Phase Ib: Dose Exploration Part-Safety | 2 years
  To assess the AEs of BC3402 in combination with durvalumab in the treatment of advanced HCC.
Phase II: Dose Expansion Part-objective response rate (ORR) | 2 years
  To assess the ORR of BC3402 in combination with durvalumab in advanced hepatocellular carcinoma (according to RECIST v1.1)

CONTACTS AND LOCATIONS:
Overall Officials: Jia Fan, MD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, China